CLINICAL TRIAL: NCT03169179
Title: Physical Activity Wearables in the Police Force: The PAW-Force Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Devon and Cornwall Police (Unknown); Dorset Police (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1617/026
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Physical Activity; Health Behavior
Keywords: Physical activity; Mobile health; Wearable fitness technology; Organisational wellness; Occupational health; Police force
MeSH Terms: conditions — Motor Activity; Health Behavior

STUDY DESIGN:
Intervention Model Description: Single group pre- and post- intervention, mixed methods exploratory trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fitbit and Bupa Boost app (Experimental): Fitbit Charge 2™ wearable physical activity monitor and Bupa Boost health and wellbeing smartphone app. 12 weeks initial use (individual goal-setting in weeks 1-6 then social features of the app in weeks 7-12) followed by a further five months of optional use (as desired by the participant).
  Interventions: Behavioral: Fitbit and Bupa Boost app

INTERVENTIONS:
Behavioral: Fitbit and Bupa Boost app — Fitbit Charge 2™ wearable physical activity monitor and Bupa Boost health and wellbeing smartphone app. 12 weeks initial use (individual goal-setting in weeks 1-6 then social features of the app in weeks 7-12) followed by a further five months of optional use (as desired by the participant).

SUMMARY:
Policing is an increasingly sedentary occupation and high levels of physical and psychological morbidities are reported by officers and staff. Wearable fitness technology may be a feasible intervention to promote physical activity and improve health.

This study aims to assess the feasibility and acceptability of introducing wearable fitness technology (Fitbit™ activity monitors linked to the 'Bupa Boost' smartphone app) as a motivator for increasing physical activity within the police force. Additional aims are to and to assess the potential impact of the intervention on physical activity, sedentary time, health and wellbeing, stress, sickness absence and self-perceived productivity, and to explore which motivational strategies (e.g. individual goal-setting vs. social competitions) are most acceptable and potentially effective and for which groups of staff.

A single-group, before and after, mixed methods exploratory trial will be conducted. Approximately 180 police officers and staff from two sites (Plymouth Basic Command Unit and North Dorset) will be recruited to take part. Participants will use the technology for 12 weeks initially followed by a further five months of optional use. A combination of questionnaire surveys, interviews and analysis of staff absence records will be used.

Data will be collected pre-intervention, mid-intervention (6 weeks), post-intervention (12 weeks) and follow-up (8 months). Primary outcomes are change in objectively recorded step count, self-reported physical activity and sedentary time. Secondary outcomes include general health and wellbeing, perceived stress and productivity, sickness absence, engagement with the intervention and perceived usability and usefulness.

This study will add to our understanding of the feasibility and acceptability of mobile fitness technology in a specific workplace setting, and inform a potential larger trial within the police force.

DETAILED DESCRIPTION:
Background:

The workplace is increasingly seen as a setting for health promotion and preventive health activities, not only to prevent occupational injury, but also to improve people's overall health and wellbeing. The police force experiences higher than average rates of illness compared to the general population, including several common risk factors for cardiovascular disease and metabolic syndrome, in addition to high stress levels. Regular physical activity plays a pivotal role in the prevention and treatment of many health-related conditions and stress reduction.

The profile of crime is changing. Lower rates of street crime and increasing rates of white collar and cybercrime mean that the act of policing is becoming a more sedentary occupation. Police officers also experience a number of barriers to undertaking physical activity including long working hours, shift work, job pressures and lack of access to training facilities.

Wearable fitness technology (smartphone applications and personal physical activity monitors) provides people with accessible ways to engage with and monitor their physical activity at their convenience. There has been a recent proliferation of research into the application of such technology for behaviour change and health improvement. However, much of this research has so far been inconclusive. For studies that have reported significant effects, these have generally been modest and short-term. Remaining knowledge gaps include which strategies should be used to maintain motivation, and the impact of the technology within different populations and subgroups.

'Bupa Boost' is a smartphone application (app) run by the private health insurer Bupa. The app is a health and wellbeing tool designed for use in the workplace, which focuses on fitness, nutrition, mindfulness and relaxation. Devon and Cornwall Police and Dorset Police will work in partnership with Bupa, which will provide the app for free to staff and support research around the app. The organisations will supply a specific activity monitor (the Fitbit Charge 2™) to synchronise with the Bupa Boost app.

Bupa Boost contains several features or strategies intended to motivate behaviour change. For the purpose of this study and based on relevant theories, the features are categorised in two 'motivational frames':

1. Individual (goal-setting to earn points and virtual rewards such as badges)
2. Social (connecting with colleagues for support and to take part in competitive and collaborative/team challenges).

Objectives and Hypotheses:

This PhD project will conduct an exploratory trial to examine the feasibility and acceptability of introducing wearable fitness technology (personal activity monitors linked to a smartphone app) as a motivator for increasing physical activity within the police force. The trial will explore engagement and acceptability of the intervention in both the short and long term, including the maintenance of physical activity behaviours.

The work will include an exploratory analysis of a range of outcomes. It is predicted that the intervention will be associated with increased levels of physical activity, which will lead to improved health and wellbeing and reduced stress of staff, and an increase in productivity and reduction in sick leave and absenteeism across the organisations.

It is hypothesised that the different motivational strategies within the app (i.e. individual and social) will appeal to different individuals. Consequently, a further aim of this study is to explore which motivational strategies (i.e. individual and social) are most acceptable and potentially effective for different groups of police staff.

Secondary objectives are to gain an understanding of the wider context of physical activity within the police force through the identification of key barriers and facilitators, to assess the feasibility and acceptability of the intervention at various levels of the organisation, and to assess the feasibility and acceptability of trial methods to inform a potential larger scale trial.

Research Questions:

1. Is the wearing of a physical activity monitor (Fitbit Charge 2™) and use of the 'Bupa Boost' app a feasible and acceptable way to increase physical activity levels within the Devon and Cornwall and Dorset police forces?
2. What is the longer term engagement and acceptability of the intervention?
3. What is the potential impact of the intervention on physical activity (and sedentary time), and are physical activity levels maintained in the longer term?
4. Do increasing levels of physical activity impact positively on health, wellbeing and stress levels within the police force?
5. Are increased levels of physical activity associated with a healthier workplace, as measured by an increase in perceived productivity and reduction in sick leave and absenteeism?
6. What is the experience and impact of the different app-based motivational strategies (individual vs. social) on the level of physical activity undertaken by police staff, and are there any differences according to age, gender or occupation?
7. What are the key facilitators and barriers to physical activity within the police force?
8. What is the perceived feasibility and acceptability of the intervention at various levels of the organisation?
9. Do the findings indicate feasibility and acceptability for a larger scale trial of wearable fitness technology within the police force?

Research Methodology:

A single group exploratory trial with a pre- and post- evaluation (i.e. before and after use of the wearable fitness technology) will be conducted. Volunteer participants from two sites, Plymouth Basic Command Unit (urban) and North Dorset (rural), will receive the intervention, i.e. the Fitbit activity monitor and Bupa Boost app.

Following an initial week of wearing the activity monitor only (for baseline data collection), participants will take part in a 12 week intervention where the activity monitor will be linked to the Bupa Boost app. They will set specific goals including increasing their step count, and they will then be encouraged to engage with all of the motivational strategies within the 'individual' frame in weeks 1-6, followed by the 'social' frame in weeks 7-12. At the end of the 12 weeks, there will be a 5 month 'maintenance phase' during which participants may continue to use the device and app if and when they desire.

Participants will be instructed to use only the device they are given (Fitbit Charge 2™) and Bupa Boost, and to use only the features that relate to the 'individual' or 'social' motivational frame as appropriate. Data on step count will be directly collected by the device; participants will send this electronically to the researcher at four different time points - pre-intervention (baseline), mid-intervention (6 weeks), post-intervention (12 weeks) and follow-up (5 months post-intervention). They will also complete a range of online questionnaires relating to their physical activity levels, health and wellbeing, stress, perceived productivity and absenteeism at the same time points.

The duration of the study will be approximately 12 months and is part of a 36 month PhD. A small pilot study will be undertaken to ensure the data collection methods are acceptable.

With participants' permission, some data will also be collected from staff occupational health records. This will include sickness and absence time, and most common reasons for sickness absence before and after the intervention.

In addition to quantitative data, there will be a parallel qualitative study to gain an understanding of participants' expectations (before the intervention) and experiences (after the intervention) of the wearable fitness technology, and facilitators of and barriers to its use and participating in physical activity. This will involve interviews with a small sample, including participants who showed various levels of engagement. There will also be a small survey with managers, commissioners and occupational health staff within the police force to assess their perceptions of the usefulness, acceptability and feasibility of the intervention.

Analysis Plan:

A pre- and post-trial analysis will be undertaken. Baseline data will be compared with post-intervention and follow-up outcomes. An appropriate statistical method (e.g. paired t-test, repeated measures analysis of variance) will be selected for the primary outcome of step count. Inferential analysis will be used for key secondary outcomes (International Physical Activity Questionnaire outcomes, SF-12 health survey, Perceived Stress Scale, absenteeism and presenteeism) where possible.

Changes in outcomes between the two motivational frames will also be compared to assess their impact, and subgroup analysis will be used to explore any potential associations between varying effectiveness and sociodemographic factors (i.e. age, gender, occupation). All statistical analyses will be performed in Stata (version 14).

All interviews will be audio-recorded and transcribed and a thematic and framework analysis will be undertaken.

Contribution and Justification of Benefit:

This research has the potential to fill some of the gaps in the existing evidence surrounding mobile fitness technology, including:

* Application of the technology to promote physical activity in a specific workplace setting;
* Identification of the preferred and potentially effective motivational/behaviour change strategies in this context;
* Sub-group differences - impact of the intervention and strategies according to age, gender and occupation;
* The study of both physical activity and sedentary behaviour (as the latter is an independent risk factor for poor health);
* Provide further insight into adherence to the use of wearable devices and mobile health technology and the longer-term impact on maintenance of physical activity

There are potential benefits to the health and wellbeing of the police force, which is likely to impact on the organisation and also the local community through the reduction of staff pressure due to sick days, increased health and wellness whilst at work and increased productivity and resilience to stress.

ELIGIBILITY:
Inclusion Criteria:

* Participants should expect to be employed within the police force for the duration of the study
* Must own (or have access to) a smartphone or tablet that is compatible with the Bupa Boost app (Apple or Android 4.0.3 or higher) with Bluetooth and internet access

Exclusion Criteria:

* Staff with severe limited mobility, who would be physically unable to increase their step count over the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Change in mean daily step count | Baseline, 6 weeks, 12 weeks, 8 months
  As recorded by the Fitbit wearable activity monitor

SECONDARY OUTCOMES:
Change in moderate to vigorous physical activity (MET-minutes per week) | Baseline, 6 weeks, 12 weeks, 8 months
  As reported in the International Physical Activity Questionnaire (IPAQ) (short form)
Change in total physical activity (MET-minutes per week) | Baseline, 6 weeks, 12 weeks, 8 months
  As reported in the International Physical Activity Questionnaire (IPAQ) (short form)
Change in weekday sedentary time (hours per day) | Baseline, 6 weeks, 12 weeks, 8 months
  As reported in the International Physical Activity Questionnaire (IPAQ) (short form)
Change in perceived health-related quality of life (physical and mental) | Baseline, 6 weeks, 12 weeks, 8 months
  From the SF-12 health survey
Change in perceived stress level | Baseline, 6 weeks, 12 weeks, 8 months
  Perceived Stress Scale 4-item version (PSS-4)
Change in personal perceived productivity | Baseline, 6 weeks, 12 weeks, 8 months
  From the absenteeism and presenteeism questions of the World Health Organisation (WHO) Health and Work Performance Questionnaire (HPQ)

OTHER OUTCOMES:
Change in sickness and absence time (including reasons for sickness absence) | Baseline through study completion (approximately 8 months)
  Objective data from occupational health records
Engagement with the intervention | 6 weeks, 12 weeks, 8 months
  Including self-reported wear time for device, usage time for app, goals set and use of app features
Perceived usability of the wearable fitness technology - questionnaire reported | 6 weeks, 12 weeks
  Ease of use as reported by participants - measured using a Likert-type 5-point rating scale
Perceived usefulness of the wearable fitness technology - questionnaire reported | 6 weeks, 12 weeks
  Usefulness/effectiveness as perceived by participants - measured using a Likert-type 5-point rating scale
Experiences of wearable fitness technology - interview reported | 6 weeks, 12 weeks, 8 months
  Semi-structured interviews will assess participant expectations and experiences of the technology, including further exploration of perceptions of usability and usefulness
Usefulness of the intervention | Approximately 12 weeks (post-intervention)
  As perceived by managers, commissioners and occupational health staff (structured interviews/survey)
Acceptability of the intervention | Approximately 12 weeks (post-intervention)
  As perceived by managers, commissioners and occupational health staff (structured interviews/survey)
Feasibility of the intervention for the wider workforce | Approximately 12 weeks (post-intervention)
  As perceived by managers, commissioners and occupational health staff (structured interviews/survey)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Buckingham, ResM, Principal Investigator — University of Exeter
Locations (2):
- United Kingdom (2):
  - Devon and Cornwall Police (Plymouth Basic Command Unit), Plymouth, Devon
  - Dorset Police (North Dorset site), Blandford Forum, Dorset

IPD SHARING:
Plan to Share IPD: No
Participants were informed that their data would be used for the purpose of this study only.

REFERENCES:
- [Derived] Buckingham SA, Morrissey K, Williams AJ, Price L, Harrison J. The Physical Activity Wearables in the Police Force (PAW-Force) study: acceptability and impact. BMC Public Health. 2020 Nov 3;20(1):1645. doi: 10.1186/s12889-020-09776-1. PMID 33143665